CLINICAL TRIAL: NCT05880745
Title: The Effect of the Level of Hand Fatigability on Multiple Sclerosis on General Fatigue and Functionality: A Controlled Study
Brief Title: The Effect of the Level of Hand Fatigability on Multiple Sclerosis on General Fatigue and Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Dudu ŞİMŞEK, MSc Physiotherapist, PhD Student,Principal Investigator, Pamukkale University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PamukkaleU-sımsek-MS-Tez-002
Record Dates: First submitted 2023-05-15; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Fatigue; Functionality; Multiple Sclerosis; Dexterity
Keywords: multiple sclerosis; fatigue; hand fatigability; manuel dexterity
MeSH Terms: conditions — Fatigue; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: age-gender matched patient and healthy groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group (Experimental): Patients with MS
  Interventions: Diagnostic Test: Nine-Hole Peg Test (NHPT)
- healthy group (Experimental): age-gender matched healthy persons
  Interventions: Diagnostic Test: Nine-Hole Peg Test (NHPT)

INTERVENTIONS:
Diagnostic Test: Nine-Hole Peg Test (NHPT) — Ataxia Rating and Rating Scale (SARA) for coordination Nine-Hole Peg Test (NHPT) and Dexterity Questionnaire-24 (DextQ-24) for manuel dexterity Beck Depression Inventory (BDI) for depression level The Fatigue Severity Scale (FSS) and Fatigue Impact Scale (FIS) for general fatigue level Static and dynamic fatigue levels for hand fatigability
  Other Names: Ataxia Rating and Rating Scale (SARA); Dexterity Questionnaire-24 (DextQ-24); Beck Depression Inventory (BDI); The Fatigue Severity Scale (FSS); Fatigue Impact Scale (FIS); Static and dynamic fatigue levels

SUMMARY:
The objective of this study is to investigate the effect of the level of hand fatigability on general fatigue and functionality by comparing Relapsing-Remitting Multiple Sclerosis individuals with age and sex-matched healthy individuals. 23 RRMS and 23 healthy people (mean age 40.08, 21 females, mean time since diagnosis 9.43 years, mean Expanded Disability Status Scale 3.23) were included in the study. To examine participants' fatigability level; for gross and pinch-grip Dynamic and Static Fatigue Index, for manual dexterity and functionality level Scale for the Assessment and Rating of Ataxia (SARA), Nine Hole Peg Test (NHPT) and Dexterity Questionnaire-24 (DextQ-24) were used. While Fatigue Severity Scale (FSS) and Fatigue Impact Scale (FIS) were used to examine general fatigue, Beck Depression Inventory (BDI) was used to assess emotional status. The mean age of healthy individuals with RRMS was 40.08 ± 9.81 years, and the EDSS means of individuals with RRMS was 3.23 ± 1.47. 21 of both groups were female and 2 were male. It was determined that the difference between MS individuals and healthy individuals' SARA, NHPT, FSS and FIS averages, initial and final strength values was statistically significant (p≤0.05), and the decrease in force in individuals with RRMS was higher than in healthy individuals. However, there was no difference between RRMS and healthy individuals in terms of fatigability levels examined with the Dynamic and Static Fatigue Index (p>0.05). While the relationship of Static and Dynamic Fatigue Index with FSS and FIS was not statistically significant, the relationship was significant with DextQ-24's dressing, daily activities and TV/CD/DVD subsections (p<0.05). In individuals with early RRMS, there is a decrease in the repetitive (dynamic) and continuous (static) contractions of the rough and pinch grip strength, and this decrease is related to the negative impact on the daily living activities and functionality of the individuals. In particular, motor fatigue should be addressed from the early stages of rehabilitation programs that will be planned to maintain the active participation of individuals with RRMS in their daily living activities. To show motor fatigue with indices, further studies with different fatigue indices and individuals with RRMS at different EDSS levels are needed.

DETAILED DESCRIPTION:
Introduction Multiple sclerosis (MS) is the most common neurological disease that causes disability in young adults. It usually progresses with exacerbations and remissions and causes various problems by affecting the central nervous system in different localizations.

Fatigue is one of the most common symptoms of MS and has the greatest impact on the patient's quality of life . Fatigability, which is defined as motor and muscle fatigue during motor tasks, is the exercise-induced decrease in the muscle's ability to produce power or force during sustainable tasks . In individuals with MS, fatigability levels are higher than in healthy individuals, as the nervous system cannot provide the necessary activation stimulus during maximum voluntary or continuous contractions . From the early stages of the disease, individuals with MS face problems such as decreased grip strength, and difficulty in holding small objects, which reduce dexterity and complicate daily living activities .

When fatigue studies in MS are examined; It was observed that the studies focused mostly on the lower extremity and walking, and the studies on the upper extremity were also quite limited . To the best of our knowledge, our study is the first in its field to evaluate rough and pinching hand fatigability, general fatigue, and functionality levels in Relapsing-Remitting MS (RRMS) patients and compare them with age- and sex-matched healthy individuals.

It is stated that the EDSS, which we use to evaluate the disability levels of RRMS patients, is not sensitive enough to evaluate functional parameters such as dexterity and cognition in MS . Therefore, other specific assessment methods such as the Ataxia Rating and Rating Scale (SARA), the Nine-Hole Peg Test (NHPT), and the Skill Questionnaire-24 (DextQ-24) were used to determine the level of functioning. SARA is an internationally accepted scale that is frequently used in the evaluation of ataxia. NHPT is the gold standard of performance-based assessment, which detects the patient's progress over time and is sensitive to changes in treatment . DextQ-24, which was developed to measure manual dexterity and consists of 24 questions, is divided into five subgroups washing/care, dressing, food and kitchen, daily activities, TV/CD/DVD. The lowest total score is 24, and the highest is 96. An increase in the score means a decrease in dexterity. Beck Depression Inventory (BDI) is a valid and reliable depression scale for neurological diseases .

The Fatigue Severity Scale (FSS) was used to determine the severity of the fatigue levels of individuals during the day, and the Fatigue Impact Scale (FIS) was used to determine the effects of fatigue on activities of daily living. The Turkish validity and reliability study of both scales was conducted by Armutlu et al. Static and dynamic fatigue levels in the coarse and pinch grip were assessed with a Jamar® digital hand dynamometer and pinch meter, respectively, in the standard measuring position recommended by the American Association of Hand Therapists . For the Dynamic Fatigue Index, a maximum of 15 voluntary contractions were requested from the participant. No rest was given between contractions and the number of remaining contractions was reported to the participant. The highest value of the first 3 contractions (MVC1) and the highest value of the last 3 contractions (MVC2) were recorded and the dynamic fatigue index was calculated with the formula 100*[1-(MVC2/MVC1)]. For the Static Fatigue Index, after a one-minute rest break, the participant was asked to maintain the maximum voluntary contraction for 30 seconds and the participant was not informed about the remaining time. Assuming that the participant can sustain the maximum voluntary contraction for 30 seconds, taking into account the area generated in the graph (Hypothetical Area Under the Force Curve [HAUC]) and the area calculated by the time the participant can walk (Actual Area Under the Power Curve [AUC]) Static Fatigue Index 100*[1- (AUC/HAUC)] formula.

The multi-dimensional evaluation of MS, which threatens all aspects of life and causes limitations in daily living activities, from the early period has an important place in the treatment and rehabilitation of individuals with MS. Determination of hand fatigability is essential to understand the decrease in performance in daily life in individuals with MS and to understand its reflection on upper extremity functionality and to plan targeted rehabilitation. Our study draws attention to the fact that hand fatigability may increase in activities that require repetitive and continuous contraction in individuals with RRMS from the early period and its relationship with upper extremity functionality. For a clearer distinction of fatigability, studies with different and more objective assessments of fatigue index and more studies with different types and different EDSS levels in individuals with RRMS are needed.

ELIGIBILITY:
Inclusion Criteria:

* Patient Group Being diagnosed with Relapsing Remitting Multiple Sclerosis. Being between the ages of 18-60. Agree to participate in the study. Not having an attack in the last 1 month. Expanded Disability Status Scale (GEDS) score between 1-5.5. Spasticity level in the wrist and finger flexors is between 0 and 1+ according to the Modified Ashworth Scale.

Not having any other neurological or orthopedic or rheumatological disease affecting the upper extremity.

Healthy Adult Group Agree to participate in the study. Being between the ages of 18-60. Not having a neurological disease or an orthopedic or rheumatological disease affecting the upper extremity.

Having similar demographic characteristics with the patient group participating in the study.

Exclusion Criteria:

* Using antidepressants. Refusal to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 1year
  determination of everyone's disease severity- high score( high disability)
Modified Ashworth Scale (MAS) | 1 year
  spacticity level range 0-5(high score increased spacticity

SECONDARY OUTCOMES:
Ataxia Rating and Rating Scale (SARA) | 1 year
  ataxia level- per item 0-2 - high score high ataxia
Nine-Hole Peg Test (NHPT), and the Dexterity Questionnaire-24 (DextQ-24) | 1 year
  manuel dexterity- min- max score 0-96- high score loss of dexterity
Beck Depression Scale | 1 year
  depression level min-max 0-63- high score high depression level
Fatigue Severity Scale (FSS) and Fatigue Impact Scale (FIS) | 1 year
  general fatigue- min -max 7-63- high score high fatigue
Dynamic and Static Fatigue Index | 1 year
  hand fatigability assessment- high score high fatigability

CONTACTS AND LOCATIONS:
Overall Officials: DUDU ŞIMŞEK, PhD student, Study Chair — Pamukkale University
Locations (1):
- Pamukkale Unıversity, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simsek D, Cetisli-Korkmaz N, Bir LS. Hand fatigability, self-reported fatigue, and functionality in individuals with multiple sclerosis: A cross-sectional study. Mult Scler Relat Disord. 2024 Nov;91:105863. doi: 10.1016/j.msard.2024.105863. Epub 2024 Sep 1. PMID 39245025

DOCUMENTS (1):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT05880745/Prot_000.pdf